CLINICAL TRIAL: NCT00762190
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized Study of the Safety of TAK-559 in the Treatment of Patients With Type 2 Diabetes Mellitus
Brief Title: Study of TAK-559 in Treating Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Hepatic safety signal identified.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-03-TL-559-016; U1111-1128-1034 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — (E)-4-(4-((5-methyl-2-phenyl-1,3-oxazol-4-yl)methoxy)benzyloxyimino)-4-phenylbutyric acid; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-559 32 mg QD + Insulin (Experimental)
  Interventions: Drug: TAK-559 and insulin
- Insulin (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: TAK-559 and insulin — TAK-559 32 mg, tablets, orally, once daily and insulin stable dose injection for up to 54 weeks.
  Arms: TAK-559 32 mg QD + Insulin
Drug: Insulin — TAK-559 placebo-matching, tablets, orally, once daily and insulin stable dose injection for up to 54 weeks.
  Arms: Insulin

SUMMARY:
The purpose of this study was to determine the safety of TAK-559, once daily (QD), in treating subjects receiving a stable dose of insulin to control type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Insulin is a primary regulator of blood glucose concentrations. A subnormal response to circulating insulin levels at target tissues leads to a decrease in insulin-mediated glucose uptake. Insulin resistance is associated with normal to high insulin levels and is often accompanied by dyslipidemia, a disruption in lipid metabolism resulting in increased triglycerides and low-density lipoprotein levels as well as decreased high-density lipoprotein levels in patients with type 2 diabetes mellitus. In the early stages of insulin resistance, a compensatory mechanism of increased insulin secretion by the pancreas maintains normal to near-normal glucose levels. Once the pancreas fails to maintain the increased insulin output, overt type 2 diabetes mellitus occurs.

Insulin also plays an important role in the metabolism of fat and proteins and exerts its influence at the peroxisome proliferator-activated receptor level. Peroxisome proliferator-activated receptor -alpha receptors are expressed predominantly in skeletal muscle, adipose tissue, heart, liver, kidney, gut, macrophages, and vascular tissue, and play a key role in energy storage, glucose homeostasis, and vascular biology. Thus, as insulin activates peroxisome proliferator-activated receptor-alpha receptors, this results in the cellular uptake of glucose. Peroxisome proliferator-activated receptor receptors are ligand-activated transcription elements that regulate gene expression necessary for metabolism. For this reason, peroxisome proliferator-activated receptors play a pivotal role in glucose homeostasis, adipocyte differentiation, and lipid storage. The genes predominantly targeted by transcription activity of activated peroxisome proliferator-activated receptor-alpha receptors are those that mediate fatty acid uptake, fatty acid oxidation, and lipoprotein metabolism. As such, peroxisome proliferator-activated receptor-alpha agonists have their greatest effect on lipid metabolism and vascular biology.

TAK-559 is a novel oxyiminoalkanoic acid under investigation for use as an oral agent in the treatment of patients with type 2 diabetes mellitus. TAK-559 has partial peroxisome proliferator-activated receptor-alpha agonist activity, potent peroxisome proliferator-activated receptor-alpha activity, and modest peroxisome proliferator-activated receptor-gamma activity at high concentrations in nonclinical models.

This study was designed to evaluate the safety of TAK-559 in the treatment of patients with type 2 diabetes mellitus who were on a stable dose of insulin.

ELIGIBILITY:
Inclusion Criteria:

* Had type 2 diabetes mellitus using American Diabetes Association diagnostic criteria, currently treated with insulin therapy.
* Required sponsor approval if older than 65 years.
* Had a Screening glycosylated hemoglobin less than or equal to 8.0%.
* Had a Screening fasting plasma glucose less than or equal to 200 mg/dL (11.1 mmol/L).
* Had a Screening low density lipoprotein less than or equal to 160 mg/dL (4.1 mmol/L).
* Had a Screening thyroid stimulating hormone level less than or equal to 5.5 μU/mL (5.5 μU/L) and greater than or equal to 0.35 μU/mL (0.35 μU/L).
* Was willing to continue dietary counseling during study and had dietary advice greater than or equal to 2.5 months prior to Screening.
* Had a Screening ejection fraction greater than or equal to 40% from echocardiogram.
* Had a Screening blood pressure less than or equal to 140/95 mm Hg.
* Was willing to perform daily self-monitoring blood glucose tests.
* A female subject of childbearing potential who was sexually active agreed to use adequate contraception, and was neither pregnant nor lactating from Screening throughout the duration of the study.
* Was in good health as determined by physician (via medical history and physical examination) other than having type 2 diabetes mellitus.
* Had clinical laboratory evaluations within normal reference range or deemed not clinically significant by the investigator or sponsor.
* Started insulin therapy at least 3 months prior to Randomization.

Exclusion Criteria:

* Had a hypersensitivity to peroxisome proliferator-activated receptor -alpha or gamma agonists, thiazolidinediones, or fibrates.
* Was diagnosed with type 1 diabetes mellitus or hemochromatosis, or had a history of ketoacidosis.
* Required greater than 2 hypertension medications to achieve adequate blood pressure control.
* Had a history of coronary angioplasty or bypass graft, or unstable angina pectoris within 1 year of Screening.
* Had a history of myocardial infarction.
* Had a history of transient ischemic attack or documented cerebrovascular accident within 6 months of Screening.
* Abdominal, thoracic, or vascular surgery within 6 months of Screening warranting exclusion (investigator's opinion).
* Had a screening creatine phosphokinase value greater than 3 times the upper limit of normal.
* Had persistent unexplained microscopic or macroscopic hematuria or history of bladder cancer.
* Had a screening triglyceride level greater than 500 mg/dL (5.6 mmol/L).
* Experienced a change in allowed lipid-lowering medication (dose or drug) within 2 months of Randomization.
* Experienced a change in blood pressure medication (dose or drug) within 1 month of Randomization.
* Had systemic corticosteroids within 1 month of Randomization.
* Had donated or received blood products within 3 months of Randomization.
* Had a condition known to invalidate glycosylated hemoglobin.
* Had a history of drug abuse or alcohol abuse within 2 years.
* Had a significant cardiovascular disease, including New York Heart Association Functional (Cardiac) Classification II, III or IV.
* Had a Screening B-Type Natriuretic Peptide greater than 100 pg/mL (100 ng/L).
* Had a history of left ventricular hypertrophy (women greater than 110 g/m2 and men greater than 134 g/m2).
* Had a clinically significant mitral insufficiency at Screening.
* Had a clinically significant aortic stenosis at Screening.
* Had a Screening body mass index greater than 45.
* Had a history of cancer with no remission within 5 years of Randomization, other than basal cell or stage 1 squamous cell carcinoma of the skin.
* Had an alanine transaminase or aspartate transaminase level greater than 3 times the upper limit of normal, active liver disease or jaundice at Screening.
* Had a positive human immunodeficiency virus, hepatitis B surface antigen, or hepatitis B e antigen test at Screening.
* Was required to take or intended to continue taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfered with the evaluation of the study medication, including:

  * oral antidiabetic agents (including sulfonylureas, alpha-glucosidase inhibitors, thiazolidinediones, peroxisome proliferator-activated receptor agonists and metformin)
  * fibrates
  * systemic corticosteroids
  * warfarin
  * rifampin
  * nicotinic acid
  * minoxidil
  * hydralazine
  * St. John's Wort
* Was participating or had participated in an investigational study within the past 30 days.
* Had a serious disease or condition at Screening or Randomization that could affect life expectancy or made it difficult to manage/follow patient according to protocol.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2003-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events. | All visits or at occurrence.
Clinical safety lab tests. | Weeks 12, 24, and Final Visit.
12-lead electrocardiogram. | Weeks: 24 and Final Visit.
Urinalysis. | Weeks: 12, 24, 36, 48 and Final Visit.
Change from Baseline in Blood pressure and pulse. | At all visits.
Change from Baseline in Body weight. | At all visits.
Left ventricular mass index by body surface area measured by echocardiogram. | Weeks: 24 and Final Visit.

SECONDARY OUTCOMES:
Change from Baseline in total daily dose of insulin. | At all visits.
Change from Baseline in triglycerides. | Weeks: 24 and Final Visit.
Change from Baseline in cholesterol. | Weeks 24 and Final Visit
Change from Baseline in total, high-density lipoproteins. | Weeks: 24 and Final Visit.
Change from Baseline in low-density lipoproteins. | Weeks 24 and Final Visit
Change from Baseline in low-density lipoprotein fractionation. | Weeks 24 and Final Visit
Change from Baseline in very low-density lipoprotein. | Weeks 24 and Final Visit
Change from Baseline in free fatty acids. | Weeks 24 and Final Visit
Change from Baseline in apolipoproteins (AI, B). | Weeks 24 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda